CLINICAL TRIAL: NCT02491710
Title: Comparison of an Inexpensive Tablet-based Laparoscopic Box Trainer With a Standard Box Trainer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Heinrich Husslein, Ass.-Prof., Staff physician, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1322/2015
Record Dates: First submitted 2015-06-27; First posted 2015-07-08 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Basic Laparoscopic Skills Training
Keywords: Surgical education; Laparoscopy; Laparoscopic suturing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-cost box trainer (Experimental): Trainees in this arm will perform their basic laparoscopic skills training on a low-cost tablet-based box trainer.
  Interventions: Device: Training on low-cost box trainer
- Standard box trainer (Active Comparator): Trainees in this arm will perform their basic laparoscopic skills training on a standard box trainer
  Interventions: Device: Training on standard box trainer

INTERVENTIONS:
Device: Training on low-cost box trainer
  Arms: Low-cost box trainer
Device: Training on standard box trainer
  Arms: Standard box trainer

SUMMARY:
Training is of great importance in laparoscopy. There are different commercially available trainers which are quite expensive and are used by trainees only inside the hospital.

The aim of this study is to find out whether basic laparoscopic skills training using an inexpensive tablet-based laparoscopic box trainer leads to equal training results (= improvement of skills) compared to practicing with a conventional commercial box trainer. Furthermore, trainee satisfaction with this home-made alternative compared to the standard trainer will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Medical students of the Medical University of Vienna

Exclusion Criteria:

* Extensive experience with laparoscopic box trainers or laparoscopic surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Fundamentals of Laparoscopy (FLS) manual Skills Score | After completion of training (4-6 weeks)

SECONDARY OUTCOMES:
Trainee satisfaction with the two different training devices | After completion of training (4-6 weeks)
  Satisfaction will be measured using a visual analogue scale (VAS)